CLINICAL TRIAL: NCT01514539
Title: Role of Ghrelin and PYY in Postpartum Body Weight Regulation and Presence in Human Milk
Brief Title: Hormonal Regulation of Postpartum Weight and Presence of Gut Peptides in Human Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Enette Larson-Meyer, Phd, RD, FACSM, University of Wyoming
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P20RR016474 (NIH)
Record Dates: First submitted 2012-01-09; First posted 2012-01-23 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Maternal Obesity Syndrome
Keywords: Human milk, Ghrelin,PYY and maternal obesity.
MeSH Terms: conditions — Pregnancy in Obesity | interventions — Cross-Sectional Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Four weeks Postpartum Lactating (Other): women between 18 and 45 who delivered their first child 4 weeks prior and who were currently lactating and planning to lactate for one year postpartum.
  Interventions: Other: cross-sectional
- Control Never Pregnant (Other): women between 18 and 45 who have never been pregnant
  Interventions: Other: cross-sectional

INTERVENTIONS:
Other: cross-sectional — Monitoring two recently discovered appetite hormones called "ghrelin" and "neuropeptide YY (PYY)." This study evaluated whether fasting or postprandial ghrelin or PYY is different btween lactating and nonlactating postpartum women matched for age, body weight, and adiposity.

SUMMARY:
Hormonal Regulation of Postpartum Weight and Presence of Gut Peptides in Human Milk Studies suggest that childbearing is an important contributor to the development of obesity in many women and that breastfeeding may be protective.

Ghrelin and peptide YY (PYY) are gut hormones involved in appetite regulation and energy homeostasis and are biological neuroendocrine signals that potentially affect body weight and adiposity/

DETAILED DESCRIPTION:
Role of Ghrelin and PYY in Postpartum Body Weight Regulation and Presence in Human Milk.

This study evaluated whether fasting or postprandial ghrelin or PYY is different between lactating and nonlactating postpartum women matched for age, body weight, and adiposity.

Eligibility Criteria: Healthy females, 18+ years old, non-smokers, no major food allergies, first-time mom, currently pregnant or within 1 month of giving birth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women (non-smokers) at least 18 years old who did not have any pregnancy complications, and gave birth to their first child within one month.
* The study is open to women who are breastfeeding or formula feeding.

Exclusion Criteria:

* Smoker,
* had twins or triples,
* had any major complication of pregnancy(example,
* gestational diabetes);
* have kidney, liver, hormonal, stomach, intestine,lung, heart or blood disease. This also includes high blood pressure;
* use prescription or over-the-counter medicine or herbal drinks or pills.
* History of depression, anxiety, disordered eating, other psychological problems, alcoholism or other substance abuse.
* Severely claustrophobic.
* Having a strong fear of needles and/or do not feel you can have blood drawn every 30 minutes from a plastic catheter.
* Are not able to or willing to fully participate in the study, and are pregnant, anemic or have a thyroid problem.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
"Role of Ghrelin and PYY in Postpartum Body Weight Regulation and Presence in Human Milk" | 5 years
  Biomedical Research Study that will provide information on reducing maternal obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Dawine E. Larson-Meyer, Phd, RD, Principal Investigator — University of Wyoming
Locations (1):
- Nutritional and Exercise Lab University of Wyoming, Laramie, Wyoming, United States